CLINICAL TRIAL: NCT02040363
Title: Impact of Exercise Training on Skeletal Muscle Capillary Maturation During Angiogenesis in COPD Patients
Brief Title: Muscle Training Induced Angiogenesis in COPD
Acronym: COPDµvasc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Montpellier (Other); 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 9224
Record Dates: First submitted 2014-01-10; First posted 2014-01-20 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Muscle Dysfunction; COPD
Keywords: COPD; skeletal muscle; angiogenesis; exercise training; intensity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- COPD Patients ~90% VO2max (Active Comparator): COPD Patients ~90% VO2max
  Interventions: Procedure: Muscular biopsy
- COPD patients ~60-65% VO2max (Active Comparator): COPD patients ~60-65% VO2max
  Interventions: Procedure: Muscular biopsy
- healthy volunteers (Placebo Comparator): healthy volunteers
  Interventions: Procedure: Muscular biopsy; Other: 5-10 weeks sport training

INTERVENTIONS:
Procedure: Muscular biopsy
Other: 5-10 weeks sport training
  Arms: healthy volunteers

SUMMARY:
COPD patients experiment a peripheral muscle dysfunction which impact their exercise tolerance and health-related quality of life. The capillary to fiber interface is reduced and impact the exercise capacity of the patients. While the muscle capillary creation in response to exercise training is blunted in COPD patients, the maturation of the neo-capillaries could also be blunted and contribute to the impaired aniogionenesis in patients. Because the capillary maturation is a sensitive and dynamic process, only different modalities of exercise training and multiple time-points of measures would allow to capture this microvascular adaptation.

Aim of the study : Compare the muscle capillary maturation in response to training at 5 and 10 weeks, in sedentary healthy subject trained at the intensity of the ventilatory threshold (60-65% of VO2max), versus :- COPD patients trained at a similar intensity (60-65% of VO2max)- COPD patients trained at a similar absolute intensity (90% of VO2max).

ELIGIBILITY:
Inclusion Criteria:

* COPD patients :
* FEV1<80%pred.
* non exacerbation during the past 4 weeks
* no oxygen therapy, -

Healthy subjects:

* <150min/week of moderate-to-vigorous physical activity,
* Voorrips score <9

Exclusion Criteria:

* Unstable comorbidity
* Long term oxygen therapy or ventilation
* Rehabilitation program during the past 12 months
* nutritional supplementation during the past 4 weeks
* allopurinol or N-acetylcystein during the past 4 weeks
* long corticosteroid treatment during the past 6 months
* hyperreactivity to xylocain
* anticoagulant or platelet aggregation inhibitors treatment
* participation to an other research study-pregnancy or impossibility to provide informed consent, ...

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Capillary-o-fiber ratio assessed by immunochemistry on a muscle biopsy of the vastus lateralis of the quadriceps | 5 weeks
Capillary-o-fiber ratio assessed by immunochemistry on a muscle biopsy of the vastus lateralis of the quadriceps | 10 weeks

SECONDARY OUTCOMES:
quadriceps endurance | 5 weeks
quadriceps endurance | 10 weeks
Pericyte coverage of skeletal muscles capillaries assessed by immunostaining of a muscle biopsy of the vastus lateralis of the quadriceps | 5 weeks
Pericyte coverage of skeletal muscles capillaries assessed by immunostaining of a muscle biopsy of the vastus lateralis of the quadriceps | 10 weeks
Effect of the serum of COPD patients and SHS on pericyte morphology and in vitro | 10 weeks
Effect of the serum of COPD patients and SHS on pericyte/endothelial cells interactions in vitro | 10 weeks
Effect of the serum of COPD patients and SHS on pericyte/endothelial cells interactions in vivo | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Farés Gouzi, Principal Investigator — University Hospital
Locations (1):
- Department of clinical Physiology - University Hospital, Montpellier, France

REFERENCES:
- [Derived] Souweine JS, Gouzi F, Badia E, Pomies P, Garrigue V, Morena M, Hayot M, Mercier J, Ayoub B, Quintrec ML, Raynaud F, Cristol JP. Skeletal Muscle Phenotype in Patients Undergoing Long-Term Hemodialysis Awaiting Kidney Transplantation. Clin J Am Soc Nephrol. 2021 Nov;16(11):1676-1685. doi: 10.2215/CJN.02390221. PMID 34750160